CLINICAL TRIAL: NCT00224003
Title: Open-Label, Multi-Center Study of the Safety and Efficacy of Ferrlecit® in the Maintenance of Iron Stores in Pediatric Hemodialysis Patients Receiving Epoetin
Brief Title: Study of the Safety and Efficacy of Ferrlecit® Maintenance Dosing in Pediatric Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Gary Hoel, RPh, PhD Executive Director, Clinical Research, Watson Laboratory, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRO2001; FDA
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-08

CONDITIONS: Anemia
Keywords: Anemia
MeSH Terms: conditions — Anemia | interventions — ferric gluconate; Sucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sodium Ferric Gluconate Complex in Sucrose.

SUMMARY:
A phase 4 clinical investigation in iron-replete pediatric hemodialysis patients, whose legal guardian had provided signed informed consent, and who had satisfied the inclusion and exclusion criteria of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric ESRD, Patients >_ 2 and <_ 16 years of age, whose legally authorized representative provided signed informed consent.
* Stabilized on chronic hemodialysis therapy with an identified need for maintenance iron therapy.
* Predetermined TSAT and serum Ferritin (at the screening visit).
* Receiving a stable EPO dosing regimen.

Exclusion Criteria:

* Receipt of any form of iron supplementation during the 2 weeks prior to the first Ferrlecit dosing.
* Hypersensitivity to Ferrlecit or any of its inactive components.
* High TSAT level.
* High Serum Ferritin

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2003-04; Primary Completion 2004-03 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hoel, RPh, PhD, Study Director — Watson Laboratories, Inc.
Locations (10):
- United States (10):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Diego, California
  - Stanford, California
  - Atlanta, Georgia
  - Boston, Massachusetts
  - Kansas City, Missouri
  - The Bronx, New York
  - Dallas, Texas
  - Seattle, Washington

REFERENCES:
- [Result] Warady BA, Zobrist RH, Finan E; Ferrlecit Pediatric Study Group. Sodium ferric gluconate complex maintenance therapy in children on hemodialysis. Pediatr Nephrol. 2006 Apr;21(4):553-60. doi: 10.1007/s00467-006-0042-5. Epub 2006 Mar 7. PMID 16520948

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Ferric Gluconate Complex
Started | 23 (First patient in: April 2, 2003)
Completed | 16 (Last patient out: March 31, 2004)
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 1
Not completed — unk | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Ferric Gluconate Complex
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13.2 (2.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Serum Ferritin
Description: Change from baseline to 2 weeks after last Fe dose
Time Frame: 14 weeks
Population: Per protocol (completer) population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Ferric Gluconate Complex
Number analyzed (Participants) | 12
ng/mL | 26.7 (240.05)

2. Secondary Outcome: Evaluate the Effect of Intravenous Administration of Ferrlecit on Hematology Parameteres, on EPO Dose, and Safety.
Time Frame: 14 weeks
Reporting Status: Not Posted

3. Primary Outcome: Transferrin Saturation
Description: Change from baseline to 2 weeks after last dose
Time Frame: 14 weeks
Population: Per protocol (completer) population
Measure: Mean (Standard Deviation); unit: %
Arm/Group | Sodium Ferric Gluconate Complex
Number analyzed (Participants) | 12
% | 2.0 (11.67)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less